CLINICAL TRIAL: NCT00002335
Title: A Phase I, Randomized, Single-Dose, Placebo-Controlled Trial to Evaluate the Safety and Pharmacokinetics of 524W91
Brief Title: The Safety and Effectiveness of 524W91
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 233A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine

SUMMARY:
To assess the safety and pharmacokinetics of single oral doses of 524W91 administered in HIV-infected patients. To determine the effects of food on bioavailability of 524W91.

DETAILED DESCRIPTION:
Patients are randomized to receive six single escalating doses of 524W91 or placebo, with each dose separated by at least a 6-day washout interval. In the time between 2 of the doses, the effect of food on pharmacokinetics will be investigated, with one dose administered in conjunction with a high-fat meal and one dose administered in a fasted state.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 count >= 200 cells/mm3.
* No active opportunistic infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy or other condition that would confound study assessment or interfere with ability to complete the study.
* Malabsorption syndrome or other gastrointestinal dysfunction that might interfere with gastrointestinal absorption.

Concurrent Medication:

Excluded on the day of each dose:

* Antiretrovirals.
* Any prescription or over-the-counter medication.
* Alcoholic beverages.
* Coffee, tea, and other xanthine-containing beverages and foods.

Patients with the following prior conditions are excluded:

History of hepatitis, pancreatitis, or cardiomyopathy within the past 5 years.

Prior Medication:

Excluded:

* Antiretrovirals within 24 hours prior to each dose.
* Any prescription or over-the-counter medications within 48 hours prior to each dose.
* Alcoholic beverages within 48 hours prior to each dose. Current alcohol or illicit drug use that may affect patient compliance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18

CONTACTS AND LOCATIONS:
Locations (1):
- ViRx Inc, San Francisco, California, United States